CLINICAL TRIAL: NCT07159594
Title: The Impact of a Weight Reduction Intervention on Clinical Outcomes in Patients With Obesity and COPD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sahlgrenska University Hospital (Other)
Collaborators: Göteborg University (Other)
Responsible Party: Principal Investigator, Jenny van Odijk, Docent, Sahlgrenska University Hospital
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SahlgrenskaUH03610
Record Dates: First submitted 2025-08-28; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: COPD; Obesity &Amp; Overweight
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Obesity; Overweight

STUDY DESIGN:
Intervention Model Description: Intervention with delayed intervention in the control arm
Masking Description: Investigator not taking part of the intervention will provide randomisation to start with diet or control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Energy restriction (Other): One arm will start as control group
  Interventions: Other: Energy restriction
- Energy restriction delayed (Other): delayed
  Interventions: Other: Energy restriction

INTERVENTIONS:
Other: Energy restriction — Diet with LED and energy restricted diet with gradually inclusion of meals
  Other Names: Energy restriction delayed

SUMMARY:
Obesity and COPD are increasingly common and often coexist, worsening health outcomes such as reduced lung function, exercise capacity, and increased systemic inflammation. While COPD was historically associated with underweight, obesity is now more prevalent among these patients and poses new challenges. Despite some evidence that weight loss may improve lung function, comprehensive interventions have not been fully studied.

The TRIO-COPD study aims to evaluate a 20-week program combining energy restriction, adequate protein intake, and structured exercise in COPD patients with obesity. The study will assess:

Primary outcome:

-Exercise capacity (6-minute walking test).

Secondary outcomes:

-Lung function (spirometry and lung volumes), -symptoms ( assessed via questionnaires), body composition (fat mass, fat-free mass, waist circumference), and inflammatory markers (e.g., IL-6, CRP, CC16).

A subgroup will also undergo sputum analysis.

The study addresses a critical gap, aiming to determine whether structured weight reduction can improve COPD symptoms, reduce inflammation, and limit muscle loss-advancing understanding of obesity's impact on COPD and providing evidence for potential treatment guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with COPD, defined by the GOLD criteria, with a forced expiratory volume in one second (FEV1) < 80% of predicted and a forced expiratory ratio of <70, with a BMI ≥ 30 kg/m2

Exclusion Criteria:

* patients with untreated cardiac disease, renal or hepatic failure, active cancer treatment, diabetes mellitus with prescribed insulin or patients with reported unintentional weight loss in the previous three months, or physical impairment that might affect the exercise capacity.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
6 minute walking test | 20 weeks

SECONDARY OUTCOMES:
Lung function | 20 weeks
  FEV₁ (Forced Expiratory Volume in 1 second)
  FVC (Forced Vital Capacity)
  FEV₁/FVC ratio

IPD SHARING:
Plan to Share IPD: Undecided
Will be added later